CLINICAL TRIAL: NCT05154760
Title: The Effectiveness of the Video Conferencing Telerehabilitation Method, Delivered in One on One and Group Sessions, in Urinary Incontinence Cases
Brief Title: Effectiveness of Video Conferencing in Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: urinary incontinence
Record Dates: First submitted 2021-09-24; First posted 2021-12-13 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2022-09

CONDITIONS: Urinary Incontinence,Stress; Telerehabilitation; Pelvic Floor Muscle Training; Videoconferencing
Keywords: urinary incontinence; tele rehabilitation; video conferencing; pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one on one video conference (Active Comparator): Pelvic floor muscle training, diaphragmatic breathing exercise, core strengthening exercise will continue for 8 weeks. Participants will be asked to practice the exercises at least 4 days in a week, and the program will be continued in the form of one on one interviews with video conference method once a week.
  Interventions: Other: Pelvic floor muscle training, diaphragmatic breathing exercise, core exercises
- group videoconference (Active Comparator): Pelvic floor muscle training, diaphragmatic breathing exercise, core strengthening exercise will continue for 8 weeks. Participants will be asked to practice the exercises at least 4 days in a week, and the program will be continued in the form of group interviews with video conference method once a week.
  Interventions: Other: Pelvic floor muscle training, diaphragmatic breathing exercise, core exercises

INTERVENTIONS:
Other: Pelvic floor muscle training, diaphragmatic breathing exercise, core exercises — An exercise program consisting of pelvic floor muscle training, diaphragmatic breathing exercise and core exercises will be applied to the patients.

SUMMARY:
Telerehabilitation (TR) refers to the provision of rehabilitation services through information and communication technologies. The most widely used of these technologies are applications such as telephone and video conferencing.

Urinary incontinence is defined as involuntary urinary incontinence ). This condition, which affects both sexes, is more common in women. Urinary incontinence is caused by dysfunction in the bladder and pelvic floor muscles in women during menopause, childbirth, or pregnancy. Urinary incontinence is a health problem that significantly affects people's social interactions, interests, and psychosocial status. It has been shown that even mild incontinence complaints cause a decrease in the quality of life in women.

Pelvic floor muscle training is one of the conservative treatment methods used in the treatment of urinary incontinence.Adding breathing exercises and deep abdominal muscle strengthening exercises to pelvic floor muscle training may be beneficial in patients with urinary incontinence.

In patients with urinary incontinence, women who are in regular communication with the supervisor during pelvic floor muscle training are more likely to gain higher from the program. However, it has not been shown that group physiotherapy is less effective than physiotherapy administered individually in reducing incontinence episodes. In the light of this information in the literature, our research hypothesis is that in patients with urinary incontinence, follow-up the pelvic floor muscle training, breathing exercise, and core exercise training with individually video conference method can have positive effects on patients' muscle strength, incontinence degree, quality of life, patient satisfaction, exercise adherence, and sexual function.

DETAILED DESCRIPTION:
During the COVID-19 pandemic in the world, telerehabilitation methods are widely used in order to ensure the continuity of patients' access to health services, as well as to reduce the likelihood of both health personnel and the patient catching the disease. Telerehabilitation (TR) refers to the provision of rehabilitation services through information and communication technologies. Information and communication technologies include secure messaging services and e-mail services, but new applications such as wearable, virtual reality and activity trackers are increasingly used in healthcare. On the other hand, real-time applications, where information is instantly exchanged between all users by telephone and video conferencing, are the most common of information and communication technologies.

Urinary incontinence is defined as the complaint of involuntary urinary incontinence. This condition, which affects both sexes, is more common in women. Urinary incontinence is caused by the disruption of the continence mechanism as a result of prostate enlargement or prostate cancer in men; In women, it is due to dysfunction in the bladder and pelvic floor muscles that occur during menopause, childbirth or pregnancy. urinary incontinence; It is classified as stress incontinence, urge incontinence, mixed type incontinence, overflow incontinence and functional incontinence. In a study conducted in our country, it was reported that stress type incontinence is the most common type of incontinence. Stress type incontinence is followed by mixed type incontinence and urge type incontinence, respectively. Urinary incontinence is a health problem that significantly affects people's social interactions, interests and psychosocial status. Studies have shown that even mild incontinence complaints cause a decrease in the quality of life in women.

Conservative treatment, pharmacological treatment and surgical interventions are used in the treatment of urinary incontinence. Pelvic floor muscle training is one of the conservative treatment methods used in the treatment of urinary incontinence. Studies in the literature have reported that pelvic floor muscle training should be included in the primary care program in women with stress or any type of incontinence, and this training causes less urinary incontinence, less urine in the pad test, and patients empty their bladders less frequently during the day. It has been shown that the pelvic floor muscles work synergistically with the diaphragm and abdominal muscles to control respiration and changes in intra-abdominal pressure. Therefore, it has been reported in the literature that adding breathing exercises and deep abdominal muscle strengthening exercises to pelvic floor muscle training in patients with urinary incontinence may be beneficial.

When the studies are examined, the programs that include pelvic floor muscle training are quite variable. Different methods were used in order to increase the effectiveness of the applied muscle training program and the adherence of the patients to the program. One of these applied methods is telerehabilitation applications. It has been shown that pelvic floor muscle training can be applied safely and effectively with telehealth applications, and significant improvements are achieved in stress incontinence and mixed type incontinence types with these applications. It has been reported that these technological methods are advantageous in order to ensure continuity of treatment without leaving the house during the pandemic process.

Women with regular contact with the supervisor during pelvic floor muscle training in patients with urinary incontinence are more likely to report their recovery. However, group physiotherapy has not been shown to be less effective than individual physiotherapy in reducing incontinence episodes. In the light of this information in the literature, pelvic floor muscle training, breathing exercise and core exercises performed individually with video conference monitoring, which is one of the telerehabilitation methods in patients with urinary incontinence, on muscle strength, incontinence degree, pelvic floor muscle thickness, symptoms on quality of life, patient satisfaction, exercise. We have established our hypothesis in terms of positive effects on commitment and sexual life. Therefore, the aim of this study is; The aim of this study is to compare the effectiveness of group video conferencing method and individual video conferencing method on urinary incontinence in patients with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 aged
* BMI 18-30 kg/m2
* Being diagnosed with stress incontinence or mixed incontinence (dominantly SUI)
* Mild or moderate incontinence (mild SUI; urinary incontinence with coughing, sneezing, laughing, or any strenuous activity. Moderate; urinary incontinence with carrying, pushing, lifting, walking, and any light physical activity)

Exclusion Criteria:

* Pregnancy
* Ongoing vulvovaginitis or urinary tract infection or malignancy
* Pelvic floor muscle strength is between 0-1 according to the Modified Oxford Scale,
* Previous surgery for SUI
* Problems with vision or inability to understand given commands
* Conservative therapy in the last 6 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Strength | Baseline
  PERFECT scheme
Pelvic Floor Muscle Strength Change | end of the 4th week
  PERFECT scheme
Pelvic Floor Muscle Strength | end of the 8th week
  PERFECT scheme
Pelvic Floor Muscle Strength change | Baseline
  Surface Electromyography
Pelvic Floor Muscle Strength change | end of the 4th week
  Surface Electromyography
Pelvic Floor Muscle Strength change | end of the 8th week
  Surface Electromyography

SECONDARY OUTCOMES:
Symptom Evaluation | Baseline
  1-h pad test: It will be used for evaluating incontinence severity. It is a test that is standardized by the International Continence Association, reveals objective results after treatment and is routinely used in incontinence clinics. At the end of the test, the weight of the pad reweighed to calculate the urinary loss. Urinary continence was defined as when the 1 h pad test less than < 2g.
Symptom Evaluation | end of the 4th week
  1-h pad test: It will be used for evaluating incontinence severity. It is a test that is standardized by the International Continence Association, reveals objective results after treatment and is routinely used in incontinence clinics. At the end of the test, the weight of the pad reweighed to calculate the urinary loss. Urinary continence was defined as when the 1 h pad test less than < 2g.
Symptom Evaluation | end of the 8th week
  1-h pad test: It will be used for evaluating incontinence severity. It is a test that is standardized by the International Continence Association, reveals objective results after treatment and is routinely used in incontinence clinics. At the end of the test, the weight of the pad reweighed to calculate the urinary loss. Urinary continence was defined as when the 1 h pad test less than < 2g.
Symptom Evaluation | Baseline
  International Consultation on Incontinence Questionnaire - Short Form (ICIQ - SF): It is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. The answers form a score ranging from 0 to 21. The higher the score, the worse the woman experiences her stress urinary incontinence to be.The overall scores can be divided into four severity categories: slight = 1-5 points, moderate = 6-12 points, severe = 13-18 points, and very severe = 19-21 points.
Symptom Evaluation | end of the 4th week
  International Consultation on Incontinence Questionnaire - Short Form (ICIQ - SF): It is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. The answers form a score ranging from 0 to 21. The higher the score, the worse the woman experiences her stress urinary incontinence to be.The overall scores can be divided into four severity categories: slight = 1-5 points, moderate = 6-12 points, severe = 13-18 points, and very severe = 19-21 points.
Symptom Evaluation | end of the 8th week
  International Consultation on Incontinence Questionnaire - Short Form (ICIQ - SF): It is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. The answers form a score ranging from 0 to 21. The higher the score, the worse the woman experiences her stress urinary incontinence to be.The overall scores can be divided into four severity categories: slight = 1-5 points, moderate = 6-12 points, severe = 13-18 points, and very severe = 19-21 points.
Symptoms Evaluation | baseline
  Urogenital Distress Inventory (UDI-6) : It will be used to evaluate the presence of different urogenital symptoms and the effect of these symptoms on the patient's quality of life. Item responses range from 0 to 3. The total score on the questionnaire is obtained by averaging the results of all items multiplied by 33 and 1/3 put scores on a scale of 0 to 100. Higher scores indicates more symptoms distress
Symptoms Evaluation | end of the 4th week
  Urogenital Distress Inventory (UDI-6) : It will be used to evaluate the presence of different urogenital symptoms and the effect of these symptoms on the patient's quality of life. Item responses range from 0 to 3. The total score on the questionnaire is obtained by averaging the results of all items multiplied by 33 and 1/3 put scores on a scale of 0 to 100. Higher scores indicates more symptoms distress
Symptoms Evaluation | end of the 8th week
  Urogenital Distress Inventory (UDI-6) : It will be used to evaluate the presence of different urogenital symptoms and the effect of these symptoms on the patient's quality of life. Item responses range from 0 to 3. The total score on the questionnaire is obtained by averaging the results of all items multiplied by 33 and 1/3 put scores on a scale of 0 to 100. Higher scores indicates more symptoms distress
Symptoms Evaluation | baseline
  Incontinence Impact Questionnaire - 7 (IIQ-7) : It will be used to evaluate the presence of different urogenital symptoms and the effect of these symptoms on the patient's quality of life, feelings and relationships. Item responses range from 0 to 3. A higher score indicates more severe symptoms and lower quality of life. The total score on the questionnaire is obtained by averaging the results of all items multiplied by 33 and 1/3 put scores on a scale of 0 to 100.
Symptoms Evaluation | end of the 4th week
  Incontinence Impact Questionnaire - 7 (IIQ-7) : It will be used to evaluate the presence of different urogenital symptoms and the effect of these symptoms on the patient's quality of life, feelings and relationships. Item responses range from 0 to 3. A higher score indicates more severe symptoms and lower quality of life. The total score on the questionnaire is obtained by averaging the results of all items multiplied by 33 and 1/3 put scores on a scale of 0 to 100.
Symptoms Evaluation | end of the 8th week
  Incontinence Impact Questionnaire - 7 (IIQ-7) : It will be used to evaluate the presence of different urogenital symptoms and the effect of these symptoms on the patient's quality of life, feelings and relationships. Item responses range from 0 to 3. A higher score indicates more severe symptoms and lower quality of life. The total score on the questionnaire is obtained by averaging the results of all items multiplied by 33 and 1/3 put scores on a scale of 0 to 100.
Symptoms Evaluation | Baseline
  Over Active Bladder -Validated 8- Question Awareness Tool (OAB-V8): It has been suggested that the questionnaire consisting of 8 questions be used as an overactive bladder screening and awareness test in patients. It is a self administered tool directed toward detecting patient suffering from over active bladder. It contains 8 items and items are measured on 6 point Likert scale. The total score range from 0 to 52 points, with a score above 8 points reflecting that the patient may have over active bladder.
Symptoms Evaluation | end of the 4th week
  Over Active Bladder -Validated 8- Question Awareness Tool (OAB-V8): It has been suggested that the questionnaire consisting of 8 questions be used as an overactive bladder screening and awareness test in patients. It is a self administered tool directed toward detecting patient suffering from over active bladder. It contains 8 items and items are measured on 6 point Likert scale. The total score range from 0 to 52 points, with a score above 8 points reflecting that the patient may have over active bladder.
Symptoms Evaluation | end of the 8th week
  Over Active Bladder -Validated 8- Question Awareness Tool (OAB-V8): It has been suggested that the questionnaire consisting of 8 questions be used as an overactive bladder screening and awareness test in patients. It is a self administered tool directed toward detecting patient suffering from over active bladder. It contains 8 items and items are measured on 6 point Likert scale. The total score range from 0 to 52 points, with a score above 8 points reflecting that the patient may have over active bladder.
Symptoms Evaluation | baseline
  Bladder diary and urination chart : The patient will be asked to record the frequency of daytime urination, the frequency of nighttime urination, the frequency of urinary incontinence for 24 hours, the frequency of the need to urinate, and the amount of fluid taken daily for the first 3 days of starting the treatment and the last 3 days before the end of the treatment.
Symptoms Evaluation | end of the 4 week
  Bladder diary and urination chart : The patient will be asked to record the frequency of daytime urination, the frequency of nighttime urination, the frequency of urinary incontinence for 24 hours, the frequency of the need to urinate, and the amount of fluid taken daily for the first 3 days of starting the treatment and the last 3 days before the end of the treatment.
Symptoms Evaluation | end of the 8 week
  Bladder diary and urination chart : The patient will be asked to record the frequency of daytime urination, the frequency of nighttime urination, the frequency of urinary incontinence for 24 hours, the frequency of the need to urinate, and the amount of fluid taken daily for the first 3 days of starting the treatment and the last 3 days before the end of the treatment.
Exercise Adherence | end of the 4th week
  Exercise adherence will be evaluated by Visual Analog Scale. The score ranges from 0 to 100. Participants will be asked to rate their degree of adherence to exercise by scoring between 0 and 100.
Exercise Adherence | end of the 8th week
  Exercise adherence will be evaluated by Visual Analog Scale. The score ranges from 0 to 100. Participants will be asked to rate their degree of adherence to exercise by scoring between 0 and 100.
Exercise Adherence | baseline
  Broome Pelvic Muscle Self-Efficacy Scale will be used for assessment of exercise adherence. It is 23-item rating scale consisting of two domains: expectations and outcome expectations.The score ranges from 0 to 100. The higher score shows more exercise adherence.
Exercise Adherence | end of the 4th week
  Broome Pelvic Muscle Self-Efficacy Scale will be used for assessment of exercise adherence. It is 23-item rating scale consisting of two domains: expectations and outcome expectations.The score ranges from 0 to 100. The higher score shows more exercise adherence.
Exercise Adherence | end of the 8 week
  Broome Pelvic Muscle Self-Efficacy Scale will be used for assessment of exercise adherence. It is 23-item rating scale consisting of two domains: expectations and outcome expectations.The score ranges from 0 to 100. The higher score shows more exercise adherence.
Patient Satisfaction | end of the 4th week
  Patient satisfaction will be evaluated by Visual analog Scale. Participants will be asked to rate their satisfaction level from the treatment by scoring between 0 and 100.
Patient Satisfaction | end of the 8th week
  Patient satisfaction will be evaluated by Visual analog Scale. Participants will be asked to rate their satisfaction level from the treatment by scoring between 0 and 100.
Sexual Function | baseline
  Female Sexual Function Scale (FSFI): It will be used for measurement of female sexual functioning during previous 4 weeks.It is a 19-item questionnaire with six dimensions. The cut off value of FSFI is 26. Lower score indicates worse sexual function.
Sexual Function | end of the 4th week
  Female Sexual Function Scale (FSFI): It will be used for measurement of female sexual functioning during previous 4 weeks.It is a 19-item questionnaire with six dimensions. The cut off value of FSFI is 26. Lower score indicates worse sexual function.
Sexual Function | end of the 8th week
  Female Sexual Function Scale (FSFI): It will be used for measurement of female sexual functioning during previous 4 weeks.It is a 19-item questionnaire with six dimensions. The cut off value of FSFI is 26. Lower score indicates worse sexual function.

CONTACTS AND LOCATIONS:
Locations (1):
- Berivan Beril Kılıç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Jul 6;3:17042. doi: 10.1038/nrdp.2017.42. PMID 28681849
- [Background] Basak T, Uzun S, Arslan F. Incontinence features, risk factors, and quality of life in Turkish women presenting at the hospital for urinary incontinence. J Wound Ostomy Continence Nurs. 2012 Jan-Feb;39(1):84-9. doi: 10.1097/WON.0b013e31823efd47. PMID 22193139
- [Background] Bezerra LO, de Oliveira MCE, da Silva Filho EM, Vicente da Silva HK, Menezes de Oliveira GF, da Silveira Goncalves AK, Pegado R, Micussi MTABC. Impact of Pelvic Floor Muscle Training Isolated and Associated with Game Therapy on Mixed Urinary Incontinence: A Randomized Controlled Trial. Games Health J. 2021 Feb;10(1):43-49. doi: 10.1089/g4h.2019.0207. Epub 2020 Jul 21. PMID 32716652
- [Background] Bo K. Pelvic floor muscle training is effective in treatment of female stress urinary incontinence, but how does it work? Int Urogynecol J Pelvic Floor Dysfunct. 2004 Mar-Apr;15(2):76-84. doi: 10.1007/s00192-004-1125-0. Epub 2004 Jan 24. PMID 15014933
- [Background] Brennan D, Tindall L, Theodoros D, Brown J, Campbell M, Christiana D, Smith D, Cason J, Lee A. A blueprint for telerehabilitation guidelines. Int J Telerehabil. 2010 Oct 27;2(2):31-4. doi: 10.5195/ijt.2010.6063. eCollection 2010 Fall. PMID 25945175
- [Background] Cacciari LP, Morin M, Mayrand MH, Tousignant M, Abrahamowicz M, Dumoulin C. Pelvic floor morphometrical and functional changes immediately after pelvic floor muscle training and at 1-year follow-up, in older incontinent women. Neurourol Urodyn. 2021 Jan;40(1):245-255. doi: 10.1002/nau.24542. Epub 2020 Oct 19. PMID 33075192
- [Background] Cam C, Sakalli M, Ay P, Cam M, Karateke A. Validation of the short forms of the incontinence impact questionnaire (IIQ-7) and the urogenital distress inventory (UDI-6) in a Turkish population. Neurourol Urodyn. 2007;26(1):129-33. doi: 10.1002/nau.20292. PMID 17083117
- [Background] Cayan S, Akbay E, Bozlu M, Canpolat B, Acar D, Ulusoy E. The prevalence of female sexual dysfunction and potential risk factors that may impair sexual function in Turkish women. Urol Int. 2004;72(1):52-7. doi: 10.1159/000075273. PMID 14730166
- [Background] Chen SY, Tzeng YL. Path analysis for adherence to pelvic floor muscle exercise among women with urinary incontinence. J Nurs Res. 2009 Jun;17(2):83-92. doi: 10.1097/JNR.0b013e3181a53e7e. PMID 19516102
- [Background] Cottrell MA, Russell TG. Telehealth for musculoskeletal physiotherapy. Musculoskelet Sci Pract. 2020 Aug;48:102193. doi: 10.1016/j.msksp.2020.102193. Epub 2020 May 30. PMID 32560876
- [Background] Çetinel B, Özkan B, Can G. ICIQ-SF Türkçe Versiyonu: Validasyon (Geçerlilik) Çalışması. Türk Üroloji Dergisi, 2004; 30: 332-8.
- [Background] Dumoulin C, Hay-Smith EJ, Mac Habee-Seguin G. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2014 May 14;(5):CD005654. doi: 10.1002/14651858.CD005654.pub3. PMID 24823491
- [Background] Grimes CL, Balk EM, Crisp CC, Antosh DD, Murphy M, Halder GE, Jeppson PC, Weber LeBrun EE, Raman S, Kim-Fine S, Iglesia C, Dieter AA, Yurteri-Kaplan L, Adam G, Meriwether KV. A guide for urogynecologic patient care utilizing telemedicine during the COVID-19 pandemic: review of existing evidence. Int Urogynecol J. 2020 Jun;31(6):1063-1089. doi: 10.1007/s00192-020-04314-4. Epub 2020 Apr 27. PMID 32342112
- [Background] Hay-Smith J, Herderschee R, Dumoulin C, Herbison P. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women: an abridged Cochrane systematic review. Eur J Phys Rehabil Med. 2012 Dec;48(4):689-705. PMID 23183454
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Hu JS, Pierre EF. Urinary Incontinence in Women: Evaluation and Management. Am Fam Physician. 2019 Sep 15;100(6):339-348. PMID 31524367
- [Background] Hui E, Lee PS, Woo J. Management of urinary incontinence in older women using videoconferencing versus conventional management: a randomized controlled trial. J Telemed Telecare. 2006;12(7):343-7. doi: 10.1258/135763306778682413. PMID 17059650
- [Background] Hung HC, Hsiao SM, Chih SY, Lin HH, Tsauo JY. An alternative intervention for urinary incontinence: retraining diaphragmatic, deep abdominal and pelvic floor muscle coordinated function. Man Ther. 2010 Jun;15(3):273-9. doi: 10.1016/j.math.2010.01.008. Epub 2010 Feb 24. PMID 20185357
- [Background] Krhut J, Gartner M, Mokris J, Horcicka L, Svabik K, Zachoval R, Martan A, Zvara P. Effect of severity of urinary incontinence on quality of life in women. Neurourol Urodyn. 2018 Aug;37(6):1925-1930. doi: 10.1002/nau.23568. Epub 2018 Mar 31. PMID 29603780
- [Background] Laycock J, Jerwood D. Pelvic floor muscle assessment: The PERFECT Scheme. Physiotherapy, 2001; 87, 631-642.
- [Background] Novara G, Checcucci E, Crestani A, Abrate A, Esperto F, Pavan N, De Nunzio C, Galfano A, Giannarini G, Gregori A, Liguori G, Bartoletti R, Porpiglia F, Scarpa RM, Simonato A, Trombetta C, Tubaro A, Ficarra V; Research Urology Network (RUN). Telehealth in Urology: A Systematic Review of the Literature. How Much Can Telemedicine Be Useful During and After the COVID-19 Pandemic? Eur Urol. 2020 Dec;78(6):786-811. doi: 10.1016/j.eururo.2020.06.025. Epub 2020 Jun 18. PMID 32616405
- [Background] Onur R, Bayrak Ö. Ürı̇ner İnkontı̇nans Tanı ve Tedavı̇. ISBN: 978-975-00112-5-2.TÜD/TÜRK Üroloji Akademisi Yayını No: 2, 2015
- [Background] Ozlu A, Yildiz N, Oztekin O. Comparison of the efficacy of perineal and intravaginal biofeedback assisted pelvic floor muscle exercises in women with urodynamic stress urinary incontinence. Neurourol Urodyn. 2017 Nov;36(8):2132-2141. doi: 10.1002/nau.23257. Epub 2017 Mar 27. PMID 28345778
- [Background] Talasz H, Kremser C, Kofler M, Kalchschmid E, Lechleitner M, Rudisch A. Phase-locked parallel movement of diaphragm and pelvic floor during breathing and coughing-a dynamic MRI investigation in healthy females. Int Urogynecol J. 2011 Jan;22(1):61-8. doi: 10.1007/s00192-010-1240-z. Epub 2010 Aug 31. PMID 20809211
- [Background] Tarcan T, Naşide M, Özgür MÖ, Akbal C. Oab V8 Aşırı Aktif Mesane Sorgulama Formu Validasyon Çalışması. Üroloji Bülteni, 2012;21, 113-116.
- [Background] Zachovajeviene B, Siupsinskas L, Zachovajevas P, Venclovas Z, Milonas D. Effect of diaphragm and abdominal muscle training on pelvic floor strength and endurance: results of a prospective randomized trial. Sci Rep. 2019 Dec 16;9(1):19192. doi: 10.1038/s41598-019-55724-4. PMID 31844133
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT05154760/Prot_SAP_001.pdf